CLINICAL TRIAL: NCT04100096
Title: A Multicenter, Randomized, Flexible-dose, Double-blind Trial of Brexpiprazole Versus Placebo for the Treatment of Adults With Borderline Personality Disorder
Brief Title: A Trial of Brexpiprazole in the Treatment of Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-201-00242
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole 2-3 Milligrams Per Day (Experimental): Participants received brexpiprazole, 2-3 milligrams per day (mg/day) tablets, orally, up to Week 12 during the treatment phase.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Participants received brexpiprazole-matching placebo tablets, orally, up to Week 12 during the treatment phase.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Tablet
  Other Names: Rexulti®
  Arms: Brexpiprazole 2-3 Milligrams Per Day
Other: Placebo — Tablet
  Arms: Placebo

SUMMARY:
There are currently no pharmacological treatments approved to treat borderline personality disorder (BPD). This trial will be conducted to evaluate the efficacy and safety of brexpiprazole for the treatment of participants diagnosed with BPD to provide a pharmacological treatment for BPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, ages 18 to 65, inclusive, at the time of informed consent
* Participants with a primary Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnosis of BPD confirmed by the Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD) at screening.
* At screening and Day 0, participants must have a total score ≥ 12 on the Zanarini Rating Scale for BPD (ZAN-BPD) scale.
* Participants who, in the investigator's judgment, require treatment with a medication for BPD.
* Participants willing to discontinue all prohibited medications to meet protocol-required washouts prior to and during the trial period.

Exclusion Criteria:

* Sexually active males or females of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of investigational medicinal product (IMP). Consensual sexual activity that cannot biologically result in pregnancy may not be participant to required birth control methods, following discussion with the medical monitor. Male participants must also agree not to donate sperm from trial screening through 30 days after the last dose of IMP.
* Women who are breastfeeding and/or who have a positive pregnancy test result prior to receiving IMP.
* Participants with a concurrent DSM-5 diagnosis of schizophrenia or schizoaffective disorder. Also, participants with a concurrent diagnosis of bipolar I disorder, bipolar II disorder, delirium, dementia, amnesia, eating disorder, antisocial personality disorder, or other cognitive disorders.
* Participants with a current diagnosis of substance or alcohol use disorder within 90 days prior to screening visit.
* Participants who fulfill the following criteria related to suicide and/or suicidal ideation are excluded:

  * Participants who have a significant risk of committing violent acts, serious self-harm, or suicide based on history or routine psychiatric status examination, or those who are homicidal or considered to be a high risk to others, or participants with a response of "yes" on the Columbia-suicide severity rating scale (C-SSRS) Suicidal Ideation Item 5, OR
  * Participants with a response of "yes" on the C-SSRS Suicidal Behavior Items, OR
  * Participants who have had 3 suicide attempts, OR,
  * Participants who have had 3 or more hospitalizations due to suicidal behavior.
* Participants who received brexpiprazole in any prior clinical trial or participants who have taken or are taking commercially available brexpiprazole (Rexulti®).
* Participants who are currently either inpatient or partially hospitalized.
* Participants who participated in a clinical trial within 90 days prior to screening or who participated in more than 2 clinical trials within a year prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (66):
  - Pillar Clinical Research, Bentonville, Arkansas
  - CI Trials, Bellflower, California
  - Care Access Research Beverly Hills, Beverly Hills, California
  - OM Research LLC, Lancaster, California
  - CalNeuro Research Group, Los Angeles, California
  - Excell Research, Oceanside, California
  - PCSD - Feighner Research, San Diego, California
  - SF-Care Inc., San Rafael, California
  - CI Trials, Santa Ana, California
  - Viking Clinical Research, Temecula, California
  - Pacific Clinical Research Management Group, Upland, California
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Institute of Living Hartford Hospital, Hartford, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Mindful Behavioral Health, Boca Raton, Florida
  - CNS Clinical Research of Coral Springs, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - New Life Medical Research Center, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Clinical Neuroscience Solutions dba CNS Healthcare, Orlando, Florida
  - APG Research, Orlando, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - The University of Chicago Hospitals, Chicago, Illinois
  - AMR Conventions Research, Naperville, Illinois
  - Neuroscience Research Institute Inc., Winfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - McLean Hospital, Belmont, Massachusetts
  - Copley Clinical, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Advanced Clinical Research Center, LLC, Bridgeton, Missouri
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates dba Midwest Research Group, Saint Charles, Missouri
  - Arch Clinical Trials LLC, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Integrative Clinical Trials, Brooklyn, New York
  - SPRI Clinical Trials LLC, Brooklyn, New York
  - Bioscience Research, LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - MindPath Care Centers, Raleigh, North Carolina
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - North Star Medical Research LLC, Middleburg Heights, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Carolina Clinical Trials Inc., Charleston, South Carolina
  - Relaro Medical Trials, LLC, Dallas, Texas
  - Earle Research, Houston, Texas
  - Red Oak Psychiatric Associates, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - The University of Texas Heath Science Center at San Antonio, San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Psychiatric Behavioral Solutions, Salt Lake City, Utah
  - Cedar Psychiatry, Springville, Utah
  - Woodstock Research Center, Woodstock, Vermont
  - Eastside Therapeutic Resource Inc dba Core Clinical Research, Everett, Washington
- Spain (6):
  - Hospital Parc Taul Parc Tauli 1, Sabadell, Barcelona
  - Institut Hospital del Mar d'Investigacions Mèdiques - IMIM, Barcelona
  - Consultoria i Projectes Sanitaris S.L. Clinic: Hestia Palau, Barcelona
  - Hospital de la Santa Creu i Sant Pau Carrer de Sant Quint, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Provincial de Zamora, Zamora
- Ukraine (5):
  - Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - Kyiv railway clinical hospital 1, Kyiv
  - Odessa Regional Medical Centre of Mental Health, Odesa
  - Communal Enterprise-Regional Institution of Mental Psychiatric Care of the Poltava Regional Council, Poltava
  - Vinnitsa National Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Rothman B, Brewer C, Chang D, Hobart M, Hefting N, McQuade RD, Grant JE. A randomised study and an extension study of brexpiprazole in patients with borderline personality disorder. Acta Neuropsychiatr. 2024 Nov 19;37:e39. doi: 10.1017/neu.2024.31. PMID 39558901
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 62 study centers in the United States, Spain, and Ukraine from 17 October 2019 to 27 Jun 2021.
Pre-assignment Details: 332 participants were enrolled out of which 324 participants were randomized to receive brexpiprazole or matching placebo in the treatment phase.
Groups:
- Brexpiprazole 2-3 Milligrams Per Day: Participants received brexpiprazole, 2-3 milligrams per day (mg/day) tablets, orally, up to Week 12 during treatment phase.
- Placebo: Participants received brexpiprazole-matching placebo tablets, orally, up to Week 12 during treatment phase.
Period: Overall Study
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Started (Started participants were those who were randomized.) | 159 | 165
Safety Population | 157 | 165
Full Analysis Set (FAS) for Enriched Participants | 112 | 111
Completed | 112 | 127
Not Completed | 47 | 38
Not completed — Adverse Event | 19 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 13 | 11
Not completed — Non-Compliance With Study Drug | 1 | 3
Not completed — Protocol Deviation | 1 | 1
Not completed — Withdrawal by Participant | 13 | 15

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants who were randomized to receive brexpiprazole or matching placebo in the treatment phase.
Groups:
- Brexpiprazole 2 to 3 Milligrams Per Day: Participants received brexpiprazole, 2-3 mg/day tablets, orally, up to Week 12 during the treatment phase.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 2 to 3 Milligrams Per Day | Placebo | Total
Number analyzed (Participants) | 159 | 165 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (10.6) | 31.0 (10.9) | 31.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 137 | 266
  Male | 30 | 28 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 19 | 22 | 41
  White | 123 | 131 | 254
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 31 | 33 | 64
  Ethnicity: Not Hispanic or Latino | 127 | 131 | 258
  Ethnicity: Unknown | 1 | 0 | 1
  Ethnicity: Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) Total Score
Description: The ZAN-BPD is a clinician-administered scale designed to assess severity of disease symptoms in participants with BPD based on clinician rating on 9 criteria. Each of the 9 criteria for BPD was rated on a 5-point anchored rating scale of 0 to 4. These scores were clustered into 4 sector scores (akin to domains) and a total score. The 4 sector scores added up to provide the overall total score for the ZAN-BPD, which ranged from 0 to 36. A higher score represented a higher severity of disease symptoms. Mixed model repeated measures = MMRM, antidepressant therapy = ADT.
Time Frame: Baseline (Day 0) to Week 10
Population: FAS for enriched participants is a subset of randomized population who met pre-defined criteria and who received at least 1 dose of double-blind investigational medicinal product (IMP) and had a baseline value and at least 1 valid post-randomization efficacy evaluation for ZAN-BPD total score. Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Brexpiprazole 2-3 Milligrams Per Day: Participants received brexpiprazole, 2-3 mg/day tablets, orally, up to Week 12 during the treatment phase.
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 86 | 91
score on a scale | -7.27 (0.80) | -6.25 (0.76)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Test type: Superiority; p = 0.2430, MMRM — Comparison was carried out using MMRM, with study center (pooled), treatment group (TG), visit, ADT status, and TG by visit interaction (BVI), gender BVI, age BVI as factors and baseline BVI as covariate. An unstructured covariance was used; Least Square (LS) Mean Difference = -1.02, 95% CI 2-sided [-2.75 to 0.70]

2. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: The severity of illness for each participant was rated using the CGI-S. CGI-S is an observer-rated scale with a total score range of 0 to 7 where a higher score represented a worse outcome. The response choices were 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline (Day 0) to Week 10
Population: FAS for enriched participants is a subset of randomized population who met pre-defined criteria and who received at least 1 valid post-randomization efficacy evaluation for ZAN-BPD total score. Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 86 | 91
score on a scale | -1.13 (0.14) | -1.09 (0.14)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Test type: Superiority; p = 0.7759, MMRM — Comparison was carried out using MMRM, with study center (pooled), TG, visit, ADT status, and TG BVI, gender BVI, age BVI as factors and baseline BVI as covariate. An unstructured covariance was used; LS Mean Difference = -0.04, 95% CI 2-sided [-0.35 to 0.27]

3. Secondary Outcome: Change From Baseline in the Patient's Global Impression of Severity (PGI-S)
Description: PGI-S is a 7-point single-item self-report scale for the participant to rate the severity of symptoms of BPD ranging from 0 to 7 where 1 denoted no symptoms and 7 denoted very severe.
Time Frame: Baseline (Day 0), Weeks 2, 4, 6, 8, 10 and 12
Population: FAS for enriched participants is a subset of randomized population who met pre-defined criteria and who received at least 1 valid post-randomization efficacy evaluation for ZAN-BPD total score. Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure. Number analyzed = number of participants with data available for analyses at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 107 | 107
score on a scale
  Change from Baseline at Week 2 | -0.33 (0.12) | -0.27 (0.12)
  Change from Baseline at Week 4: number analyzed (Participants) | 105 | 106
  Change from Baseline at Week 4 | -0.60 (0.15) | -0.35 (0.14)
  Change from Baseline at Week 6: number analyzed (Participants) | 97 | 95
  Change from Baseline at Week 6 | -0.91 (0.15) | -0.72 (0.14)
  Change from Baseline at Week 8: number analyzed (Participants) | 93 | 91
  Change from Baseline at Week 8 | -0.99 (0.14) | -0.69 (0.14)
  Change from Baseline at Week 10: number analyzed (Participants) | 86 | 88
  Change from Baseline at Week 10 | -0.90 (0.15) | -0.79 (0.14)
  Change from Baseline at Week 12: number analyzed (Participants) | 76 | 84
  Change from Baseline at Week 12 | -1.00 (0.16) | -0.86 (0.15)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 2; Test type: Superiority; p = 0.6585, MMRM — Derived from an MMRM with fixed effects of treatment, (pooled) trial site, visit, ADT status (with/without background ADT), treatment BVI, gender BVI, covariates of baseline BVI and age BVI; LS Mean Difference = -0.06, 95% CI 2-sided [-0.32 to 0.20] — Derived from an MMRM with fixed effects of treatment, (pooled) trial site, visit, ADT status (with/without background ADT), treatment BVI, gender BVI, covariates of baseline BVI and age BVI
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 4; Test type: Superiority; p = 0.1181, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.25, 95% CI 2-sided [-0.57 to 0.06] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.2431, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.19, 95% CI 2-sided [-0.51 to 0.13] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 8; Test type: Superiority; p = 0.0638, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.30, 95% CI 2-sided [-0.61 to 0.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 10; Test type: Superiority; p = 0.5050, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.11, 95% CI 2-sided [-0.44 to 0.22] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.4277, MMRM — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -0.14, 95% CI 2-sided [-0.48 to 0.21] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Patient's Global Impression of Change (PGI-C) Scale Score
Description: A 7-point single-item self-report scale depicting a participant's rating of overall change in their condition since starting trial medication. Participants answered the question: "Since starting study medication, how much have their symptoms of Borderline Personality Disorder changed?" with a score ranging from 1 to 7 where 1 denoted very much improved and 7 denoted very much worse.
Time Frame: Weeks 2, 4, 6, 8,10 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 109 | 110
score on a scale
  Week 2: number analyzed (Participants) | 108 | 109
  Week 2 | 3.38 (0.89) | 3.30 (0.93)
  Week 4 | 3.23 (1.26) | 3.25 (1.22)
  Week 6 | 2.94 (1.14) | 3.15 (1.11)
  Week 8 | 2.94 (1.10) | 3.11 (1.12)
  Week 10 | 2.89 (1.26) | 2.97 (1.20)
  Week 12 | 2.88 (1.19) | 2.96 (1.14)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 2; Test type: Superiority; p = 0.6225, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the Cochran-Mantel-Haenszel (CMH) Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.18 to 0.30] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 4; Test type: Superiority; p = 0.9145, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.35 to 0.31] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 3: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.1535, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.52 to 0.08] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 4: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 8; Test type: Superiority; p = 0.1922, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.50 to 0.10] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 5: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 10; Test type: Superiority; p = 0.6488, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.40 to 0.25] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 6: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.5992, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.40 to 0.23] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site

5. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Scale Score
Description: Participant's condition was assessed using CGI-I scale. CGI-I is an observer-rated scale with a total score of 0 to 7 and a higher score represents a worse outcome. The score included the following response choices: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Weeks 2, 4, 6, 8, 10 and 12
Population: FAS for enriched participants is a subset of randomized population who met pre-defined criteria and who received at least 1 valid post-randomization efficacy evaluation for ZAN-BPD total score. Number analyzed = number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 110 | 110
score on a scale
  Week 2: number analyzed (Participants) | 110 | 109
  Week 2 | 2.99 (0.96) | 2.99 (0.97)
  Week 4 | 2.89 (1.04) | 3.00 (1.20)
  Week 6 | 2.62 (1.05) | 2.77 (1.21)
  Week 8 | 2.39 (1.06) | 2.79 (1.26)
  Week 10 | 2.45 (1.18) | 2.61 (1.20)
  Week 12 | 2.37 (1.19) | 2.65 (1.17)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 2; Test type: Superiority; p = 0.6579, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.29 to 0.19] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 4; Test type: Superiority; p = 0.3728, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.43 to 0.16] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 3: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.1684, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.50 to 0.09] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 4: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 8; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.74 to -0.13] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 5: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 10; Test type: Superiority; p = 0.2087, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.51 to 0.11] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site
Statistical Analysis 6: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.0389, Cochran-Mantel-Haenszel — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.64 to -0.02] — Comparison between TGs was carried out using the CMH Row Mean Score Differ Test controlling for trial site

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant administered an IMP and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE that started after start of study treatment.
Time Frame: From Baseline (Day 0) to 21 days after last dose (Up to Week 15)
Population: Safety population (SP) included those participants who received at least 1 dose of study drug (brexpiprazole or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 157 | 165
Participants | 95 | 79

7. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Test Values
Description: Laboratory parameters included hematology(Hem), serum chemistry(Che) and urinalysis(Uri). Criterion:Che-Alkaline Phosphatase (Units/liter [U/L]):≥3 x ULN, Aspartate Aminotransferase (U/L):≥3 x ULN,Bilirubin (mg/deciliter[dL]):≥2.0,Cholesterol(Cho);Cho,fasting(mg/dl):≥240,Creatine Kinase(U/L):≥3 x ULN, Creatinine(mg/dL):≥2.0,Glucose (Glu);Glu,fasting(mg/dL):100,High Density Lipoprotein (HDL) Cho (mg/dL):Male (M) < 40or Female (F) <50, Low Density Lipoprotein (LDL) Cho(mg/dL):≥160,Prolactin (nanograms/milliliter [ng/mL]):>1 x ULN,Triglyceride (mg/dL):≥150,Urate(mg/dL): M ≥10.5 or F ≥8.5,Urea Nitrogen (mg/dL):≥30,Hem-Eosinophils (Eosi) (10^9 L):≥10%,Hematocrit (%): M ≤37% and ≥3 percentage (per) point decrease from baseline or F≤32% and ≥3per point decrease from baseline, Hemaglobin(gram per deciliter [g/dL]):M ≤11.5 or F ≤9.5,Leukocytes(10^9/L):≤2.8 x10^3/uL,≤16.0 x10^3/uL,Platelets(10^9/L):≤75 x10^3/ uL,≥700 x10^3/uL,Uri-Glu,urine; Protein,urine:Increase of ≥2U.
Time Frame: From first dose of study drug up to Week 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Only those categories with at least one participant with event are reported. Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure. Number analyzed = total number of participants with at least one post-baseline numeric result for given laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 146 | 157
Participants
  Che: Alkaline Phosphatase, High | 1 | 0
  Che: Aspartate Aminotransferase, High: number analyzed (Participants) | 146 | 156
  Che: Aspartate Aminotransferase, High | 1 | 0
  Che: Bilirubin, High: number analyzed (Participants) | 137 | 150
  Che: Bilirubin, High | 0 | 2
  Che: Cho, High: number analyzed (Participants) | 55 | 56
  Che: Cho, High | 2 | 4
  Che: Cho Fasting, High: number analyzed (Participants) | 118 | 129
  Che: Cho Fasting, High | 13 | 7
  Che: Creatine Kinase, High | 4 | 3
  Che: Creatinine, High | 1 | 0
  Che: Glu Fasting, High: number analyzed (Participants) | 119 | 130
  Che: Glu Fasting, High | 29 | 30
  Che: HDL Cho, Fasting, Low: number analyzed (Participants) | 118 | 129
  Che: HDL Cho, Fasting, Low | 46 | 42
  Che: Low LDL Cho, High: number analyzed (Participants) | 55 | 56
  Che: Low LDL Cho, High | 3 | 4
  Che: LDL Cholesterol, Fasting, High: number analyzed (Participants) | 118 | 129
  Che: LDL Cholesterol, Fasting, High | 11 | 8
  Che: Prolactin, High: number analyzed (Participants) | 130 | 143
  Che: Prolactin, High | 41 | 7
  Che: Triglyceride, Fasting, High: number analyzed (Participants) | 118 | 129
  Che: Triglyceride, Fasting, High | 35 | 25
  Che: Urate, High | 1 | 0
  Che: Urea Nitrogen, High | 2 | 0
  Hem: Eosi/Leukocytes Ratio, High: number analyzed (Participants) | 146 | 154
  Hem: Eosi/Leukocytes Ratio, High | 4 | 2
  Hem: Hematocrit, Low: number analyzed (Participants) | 146 | 153
  Hem: Hematocrit, Low | 2 | 4
  Hem: Hemoglobin, Low: number analyzed (Participants) | 146 | 154
  Hem: Hemoglobin, Low | 2 | 2
  Hematology: Leukocytes, Low: number analyzed (Participants) | 146 | 154
  Hematology: Leukocytes, Low | 0 | 1
  Hem: Leukocytes, High: number analyzed (Participants) | 146 | 154
  Hem: Leukocytes, High | 2 | 0
  Hem: Platelets, Low: number analyzed (Participants) | 146 | 154
  Hem: Platelets, Low | 0 | 2
  Uri: Glu, Urine, High | 0 | 1
  Uri: Protein, Urine, High | 1 | 0

8. Secondary Outcome: Number of Participants With Potential Clinical Relevant Laboratory Test Values - Prolactin
Description: New onset (> 1 x upper limit of normal {ULN}, > 2 x ULN, 3 X ULN) prolactin means a participant who attains a categorical change during treatment phase but not at baseline. Only those categories with at least one participant with event are reported.
Time Frame: Week 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 130 | 143
Participants
  Prolactin: >1 x ULN | 37 | 4
  Prolactin: >2 x ULN | 1 | 1

9. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Abnormalities in Vital Signs
Description: Vital Signs included orthostatic hypotension, heart rate (HR), systolic and diastolic blood pressure (bp), and weight. Potential clinical relevance criterion: Orthostatic Hypotension:>= 20 millimeters of mercury (mmhg) decrease in systolic bp and >= 25 beats per minute (bpm) increase in HR from supine to standing; HR Standing (bpm):< 50 and decrease >= 15,> 120 and increase >= 15; HR Supine (bpm): < 50 and decrease >= 15,>120 and increase >= 15; Systolic BP Standing (mmhg):< 90 and decrease >=20,> 180 and increase >= 20; Systolic BP Supine (mmhg):< 90 and decrease >= 20, >180 and increase >= 20; Diastolic BP Standing (mmHg): < 50 and decrease >= 15,> 105 and increase >= 15; Diastolic BP Supine (mmHg):< 50 and decrease >= 15, > 105 and increase >= 15; Weight (kilograms[kg]): Decrease or increase >= 7%. Only those categories with at least one participant with event are reported.
Time Frame: From first dose of study drug up to Week 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed = number of participants with data available for analyses for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 154 | 165
Participants
  Orthostatic Hypotension: Low | 0 | 1
  Heart Rate Standing, High | 2 | 0
  Heart Rate Supine, Low | 1 | 1
  Systolic Blood Pressure Standing, Low | 1 | 1
  Systolic Blood Pressure Supine, Low | 1 | 0
  Weight, Increase | 5 | 3
  Weight, Decrease | 25 | 12

10. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline (Day 0), Weeks 2, 4, 6, 8, 10, and 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed = number of participants with data available for analyses for this outcome measure. Number analyzed = number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 154 | 165
kilogram (kg)
  Baseline (Day 0) | 78.60 (22.15) | 78.85 (22.33)
  Change From Baseline at Week 2: number analyzed (Participants) | 145 | 155
  Change From Baseline at Week 2 | 0.27 (1.15) | 0.09 (1.62)
  Change From Baseline at Week 4: number analyzed (Participants) | 136 | 143
  Change From Baseline at Week 4 | 1.05 (1.92) | -0.05 (2.02)
  Change From Baseline at Week 6: number analyzed (Participants) | 125 | 133
  Change From Baseline at Week 6 | 1.39 (2.25) | 0.20 (2.21)
  Change From Baseline at Week 8: number analyzed (Participants) | 117 | 131
  Change From Baseline at Week 8 | 1.55 (2.75) | -0.03 (2.41)
  Change From Baseline at Week 10: number analyzed (Participants) | 111 | 125
  Change From Baseline at Week 10 | 2.09 (2.96) | 0.37 (2.72)
  Change From Baseline at Week 12: number analyzed (Participants) | 109 | 124
  Change From Baseline at Week 12 | 1.74 (3.09) | 0.30 (2.75)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 2; Test type: Superiority; p = 0.2720, ANCOVA — ANCOVA model, with treatment as main effect and baseline value as covariate, is used for change from baseline of case comparisons; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.14 to 0.50]
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 4; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [0.63 to 1.56]
Statistical Analysis 3: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.63 to 1.73]
Statistical Analysis 4: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 8; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 1.57, 95% CI 2-sided [0.92 to 2.21]
Statistical Analysis 5: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 10; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [0.99 to 2.45]
Statistical Analysis 6: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [0.68 to 2.19]

11. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Baseline (Screening: Day -21 to Day -1), Week 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed= number of participants with data available for analyses for this outcome measure. Number analyzed= number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 134 | 146
centimeter
  Baseline (Screening: Day -21 to Day -1) | 89.74 (17.54) | 90.01 (17.25)
  Change from Baseline at Week 12: number analyzed (Participants) | 109 | 124
  Change from Baseline at Week 12 | 1.07 (5.23) | -0.32 (5.76)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.0620, ANCOVA; ANCOVA model, with treatment as main effect and baseline value as covariate, is used for change from baseline of case comparisons; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-0.07 to 2.68]

12. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: BMI is defined as weight in kilograms divided by the square of height in meters.
Time Frame: Baseline (Day 0), Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 154 | 165
kilograms per square meter (kg/m^2)
  Baseline (Day 0) | 27.35 (7.49) | 28.52 (7.69)
  Change From Baseline at Week 2: number analyzed (Participants) | 145 | 155
  Change From Baseline at Week 2 | 0.09 (0.42) | 0.05 (0.62)
  Change From Baseline at Week 4: number analyzed (Participants) | 136 | 143
  Change From Baseline at Week 4 | 0.38 (0.68) | -0.00 (0.75)
  Change From Baseline at Week 6: number analyzed (Participants) | 125 | 133
  Change From Baseline at Week 6 | 0.50 (0.81) | 0.09 (0.83)
  Change From Baseline at Week 8: number analyzed (Participants) | 117 | 131
  Change From Baseline at Week 8 | 0.57 (1.01) | 0.00 (0.89)
  Change From Baseline at Week 10: number analyzed (Participants) | 111 | 125
  Change From Baseline at Week 10 | 0.76 (1.10) | 0.15 (1.00)
  Change From Baseline at Week 12: number analyzed (Participants) | 109 | 124
  Change From Baseline at Week 12 | 0.64 (1.17) | 0.13 (1.01)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 2; Test type: Superiority; p = 0.4613, ANCOVA; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.08 to 0.17]
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 4; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.21 to 0.55]
Statistical Analysis 3: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.0001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.21 to 0.61]
Statistical Analysis 4: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 8; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [0.33 to 0.80]
Statistical Analysis 5: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 10; Test type: Superiority; p = 0, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [0.34 to 0.88]
Statistical Analysis 6: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.0004, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.23 to 0.80]

13. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Abnormalities in 12-Lead Electrocardiogram (ECG) Parameters
Description: ECG parameters analyzed included rhythm, conduction and ST/T morphology. Potential clinical relevance criterion: Rhythm- Supraventricular Premature Beat: not present at baseline and present post baseline, Ventricular Premature Beat: not present at baseline and present post baseline, Conduction- Right Bundle Branch Block: not present at baseline and present post baseline, ST/T Morphology- Symmetrical (Sym) T-Wave Inversion: not present at baseline and present post baseline. Only those categories with at least one participant with event are reported.
Time Frame: Week 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed= number of participants with data available for analyses for this outcome measure. Number analyzed = total number of participants with at least one post-baseline numeric result for the given ECG parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 133 | 143
Participants
  Rhythm: Supraventricular Premature Beat: number analyzed (Participants) | 131 | 141
  Rhythm: Supraventricular Premature Beat | 0 | 1
  Rhythm: Ventricular Premature Beat: number analyzed (Participants) | 133 | 141
  Rhythm: Ventricular Premature Beat | 1 | 0
  Conduction: Right Bundle Branch Block | 1 | 0
  ST/T Morphology: Symmetrical T-Wave Inversion | 0 | 1

14. Secondary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS consisted of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item was rated on a 5-point scale, with a score of zero representing the absence of symptoms and a score of 4 representing a severe condition. The SAS total score was the sum of the scores for all 10 items and ranged from 0 to 40. Higher scores indicated worst outcome.
Time Frame: Baseline (Day 0), Week 6 and 12
Population: SP: Participants who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure. Number analyzed = number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 138 | 148
score on a scale
  Baseline (Day 0) | 0.18 (0.65) | 0.24 (0.92)
  Change from Baseline at Week 6: number analyzed (Participants) | 123 | 133
  Change from Baseline at Week 6 | 0.04 (0.76) | -0.08 (0.55)
  Change from Baseline at Week 12: number analyzed (Participants) | 105 | 122
  Change from Baseline at Week 12 | 0.04 (0.88) | -0.05 (0.63)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.1687, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.04 to 0.25]
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.1874, ANCOVA — Analysis of covariance (ANCOVA) model, with treatment as main effect and baseline value as covariate, is used for change from baseline of case comparisons; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.06 to 0.29]

15. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: AIMS assessment consisted of 10 items describing symptoms of dyskinesia (muscles of facial expression, lips and perioral area, jaw, tongue, upper extremities, lower extremities, neck/shoulders/hips, overall movement severity, incapacitation, participant awareness). Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) were observed unobtrusively while participant was at rest (e.g., in waiting room), and study physician would make global judgments on participant's dyskinesia's (items 8 through 10). Each item was rated on 5-point scale of severity from 0 (none) to 4 (severe) and assessment of problems with teeth or dentures (yes = 1, no = 0) and if the participant normally wears dentures (yes = 1, no = 0). Total score ranged from 0 to 42. Higher scores indicated worst outcome.
Time Frame: Baseline (Day 0), Weeks 6 and 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 142 | 148
score on a scale
  Baseline (Day 0) | 0.03 (0.20) | 0.04 (0.42)
  Change from Baseline at Week 6: number analyzed (Participants) | 128 | 136
  Change from Baseline at Week 6 | -0.02 (0.25) | 0.09 (0.87)
  Change from Baseline at Week 12: number analyzed (Participants) | 108 | 124
  Change from Baseline at Week 12 | -0.02 (0.27) | 0.07 (0.73)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.0974, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.25 to 0.02]
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.3910, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.20 to 0.08]

16. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS): Global Clinical Assessment of Akathisia Score
Description: The BARS consisted of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The global clinical evaluation was made on a 6-point scale, with zero representing absence of symptoms and a score of 5 representing severe akathisia.
Time Frame: Baseline (Day 0), Weeks 6 and 12
Population: Safety population included those participants in who received at least 1 dose of study drug (brexpiprazole or placebo). Overall number of participants analyzed = number of participants with data available for analysis for this outcome measure. Number analyzed = number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 142 | 149
score on a scale
  Baseline (Day 0) | 0.08 (0.27) | 0.12 (0.40)
  Change from Baseline at Week 6: number analyzed (Participants) | 129 | 136
  Change from Baseline at Week 6 | 0.15 (0.59) | -0.04 (0.37)
  Change from Baseline at Week 12: number analyzed (Participants) | 108 | 125
  Change from Baseline at Week 12 | 0.06 (0.53) | -0.05 (0.33)
Statistical Analysis 1: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 6; Test type: Superiority; p = 0.0063, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.15, 9% CI 2-sided [0.04 to 0.26]
Statistical Analysis 2: Comparison: Brexpiprazole 2-3 Milligrams Per Day vs Placebo; Week 12; Test type: Superiority; p = 0.0670, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.01 to 0.19]

17. Secondary Outcome: Number of Participants With Suicidal Behavior and Suicidal Ideation As Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was monitored using the C-SSRS. Suicidality was defined as at least one occurrence of suicidal ideation (including wish to be dead, non-specific suicidal thought, suicidal ideation-no intent, ideation with intent, no plan, ideation with plan/intent) or at least one occurrence of suicidal behavior (actual attempt, non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts/behavior, suicidal behavior) for the assessment period.
Time Frame: Baseline (Day 0) to Week 12
Population: Safety population included those participants who received at least 1 dose of study drug (brexpiprazole or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
Number analyzed (Participants) | 157 | 165
Participants
  Suicidal Behavior | 42 | 29
  Suicidal Ideation | 78 | 70

ADVERSE EVENTS:
Time Frame: From Baseline (Day 0) to 21 days after last dose (up to Week 15)
Description: Safety population included randomized participants who received at least 1 dose of study drug (brexpiprazole or placebo).
Arm/Group | Brexpiprazole 2-3 Milligrams Per Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/165
Serious Adverse Events (participants affected / at risk) | 5/157 | 2/165
Other Adverse Events (participants affected / at risk) | 69/157 | 45/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2-3 Milligrams Per Day (N=157) | Placebo (N=165)
Gastritis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Dissociation (Psychiatric disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2-3 Milligrams Per Day (N=157) | Placebo (N=165)
Fatigue (General disorders) | 12 | 6
Weight Increased (Investigations) | 10 | 4
Increased Appetite (Metabolism and nutrition disorders) | 8 | 4
Akathisia (Nervous system disorders) | 22 | 2
Headache (Nervous system disorders) | 8 | 12
Somnolence (Nervous system disorders) | 8 | 5
Anxiety (Psychiatric disorders) | 13 | 9
Insomnia (Psychiatric disorders) | 15 | 10
Restlessness (Psychiatric disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT04100096/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04100096/SAP_001.pdf